CLINICAL TRIAL: NCT04716400
Title: A Cluster Randomized Controlled Trial of the Intervention "Stop Sexual Harassment" in Norwegian Secondary Schools
Brief Title: Effectiveness Study of the Intervention "Stop Sexual Harassment" in Secondary School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: University of Bergen (Other); Boston College (Other); Norwegian Council for Mental Health (Other); The Dam Foundation (Other)
Responsible Party: Principal Investigator, Hilde Slåtten, Researcher 2, NORCE Norwegian Research Centre AS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NORCE; Funder (Other: Dam Foundation)
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Sexual Harassment; Anti-Gay Bias; Non Sexual Harassment; Gender-based Violence; Gender Bias; Bullying; Aggression; Depressive Symptoms; Anxiety; Mental Health
Keywords: Sexual harassment; Gendered harassment; Homophobic harassment; Intervention program; RCT study; Secondary school; Youth; Teachers; Pupils; LGBTQ
MeSH Terms: conditions — Sexual Harassment; Homophobia; Harassment, Non-Sexual; Sexism; Bullying; Aggression; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled study. The randomization is at school level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): "Stop sexual harassment"
  Interventions: Behavioral: Stop sexual harassment
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Stop sexual harassment — Teachers will be introduced to a digital course on the prevention of sexual- and gendered harassment. In the course they will provided with a manual containing eight lessons to be held for the pupils. Each lesson will last 45 minutes and consist of a short lecture and practical activities for the pupils.
  Arms: Intervention group

SUMMARY:
"Stop sexual harassment" is a school based intervention tailored to reduce sexual- and gendered harassment among pupils in secondary school. The first aim of this study is to test to what extent "Stop sexual harassment" reduces sexual harassment and harassment based on sexual orientation and gender expression (gendered harassment) among 8th to 10th grade pupils in secondary school. The second aim of the study is to test to what extent the intervention increases teachers' responses to sexual- and gendered harassment among pupils. The intervention consists of eight lessons which address the prevention of sexual- and gendered harassment.

METHOD: A minimum 32 schools with at least 3840 pupils will participate in a cluster randomized controlled trial. Participating schools will be randomly assigned to intervention schools and control schools. At the intervention schools, teachers will be introduced to "Stop sexual harassment" through a digital course which will provide them with a manual containing eight lessons to be held for the pupils. At the control schools there will not be any intervention. The effects of the intervention on pupils will be determined by assessing their experiences with sexual and gendered harassment, and internalized and externalized problems prior to the intervention (T1), shortly after the intervention (T2) and six moths after the intervention (T3). The effects of the intervention on teachers will be determined by assessing the teachers' experiences of responding to sexual and gendered harassment among pupils.

HYPOTHESIS: It is expected that the intervention "Stop sexual harassment" will lead to reduced sexual and gendered harassment perpetration and victimization, and less internalized and externalized problems among the pupils in secondary school, and that teachers will more frequently take action when sexual- and gendered harassment is encountered among the pupils.

DETAILED DESCRIPTION:
AIMS AND HYPOTHESIS The first aim of this study is to test the effects of "Stop sexual harassment", a sexual- and gendered harassment prevention intervention in secondary school among 8th to 10th grade pupils. The second aim of the study is to test the effects of the intervention on teachers' responses to sexual- and gendered harassment among the pupils. "Stop sexual harassment" is targeted at both pupils and teachers with the intention of reducing sexual harassment and harassment based on sexual orientation and gender expression (gendered harassment) among the pupils. It is hypothesized that the intervention will lead to reduced sexual- and gendered harassment perpetration and victimization and less internalized and externalized problems among the pupils. It is also hypothesized that the intervention will lead to teachers more frequently taking action when sexual- and gendered harassment is encountered among pupils.

DESIGN AND METHOD Recruitment: All secondary schools (8th to 10th grade) in three counties (Vestland, Nordland and former county Buskerud) in Norway will be invited to take part in the intervention.

Design: A cluster randomized controlled trial will be used to test the effects of the intervention. Participating schools will be randomly assigned to intervention schools and control schools.

Assessment: Questionnaires will be administered to pupils and teachers, prior to the intervention to obtain a baseline level (T1), shortly after the intervention (T2), and about six months after the intervention (T3). Previously tested instruments to assess to what extent the intervention leads to reduction in sexual harassment and harassment based on sexual orientation and gender expression among the pupils will be utilized. Teachers' responses to the pupils' sexual and gendered harassment will also be assessed.

Data analytic plan and power analysis: The data will be analyzed with both simple descriptive (such as correlations, frequency tables) and advanced statistical methods. With regard to the latter, 3 level multilevel modelling will be used to assess the impact of the intervention on the outcome variables. Multilevel modelling takes into account the hierarchical design of the data due to cluster randomization by school (level 3) and school class (level 2). Cluster effects were approximated (Intra Class Correlation; ICC) influencing the main outcomes (Sexual harassment, emotional problems, attitudes towards homosexuals) by taking advantage of data from previous studies. These studies indicate that whereas relatively little (often less than 5%) of the total variance of sexual harassment victimization, bullying and emotional problems are at the school and/or school class level, a still limited amount of studies suggests that this might not be the case for instance attitudes towards homosexuals where as much as 12,5 - 30% of the total variance have been explained by school/class levels. Power calculations, by the use the Optimal Design Software, showed that with a .05 level of significance, power = .80, ICC level 2 = .25, ICC level 3=0.05, number of cluster level 2=6 (classes) with a cluster size=20 (pupils), 38 schools are needed to be able to detect effect sizes of .30 (about medium effects according to Cohen (1988). The power of the analyses can be increased by including the pre-intervention measure of the outcome variable. Assuming the average school level of the outcome variable at pre-intervention explains 50 or 30 percent of the variation of the outcome variable at post-test, decreases the number of schools to 30 and 32, respectively, given the same assumptions as above. It was therefore decided to include at least 32 schools (16 intervention schools) to guard against the possibility of type II errors. A minimum of 3840 pupils will thus take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pupils belonging to classes where their main teacher has agreed to participate in the intervention

Exclusion Criteria:

* Is not able to read and write a minimum level of Norwegian

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2037 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline sexual harassment | Two months
  Experiences of sexual harassment in schools (AAUW, 2001; 2011)
Change from baseline sexual harassment at eight months | Two months
  Experiences of sexual harassment in schools (AAUW, 2001; 2011)
Change from baseline sexual harassment at one year | Two months
  Experiences of sexual harassment in schools (AAUW, 2001; 2011)
Baseline gendered harassment | Two months
  Experiences of homophobic harassment, and harassment due to sexual orientation and gender non-conformity (Martin-Storey & August, 2016; Poteat, 2014)
Change from baseline gendered harassment at eight months | Two months
  Experiences of homophobic harassment, and harassment due to sexual orientation and gender non-conformity (Martin-Storey & August, 2016; Poteat, 2014)
Change from baseline gendered harassment at one year | Two months
  Experiences of homophobic harassment, and harassment due to sexual orientation and gender non-conformity (Martin-Storey & August, 2016; Poteat, 2014)

SECONDARY OUTCOMES:
Baseline internalized problems | Two months
  Moods and Feelings Questionnaire (Angold, 1995; Larson, Ingul, Jozefiak, Leikanger & Sund, 2016; Lundervold, Brevik, Possserud, Stormark & Hysing, 2013). Screen for Child Anxiety Related Disorders (Birmaher, Khetarpal, Cully, Brent &McKenzie, 1996)
Change from internalized problems at eight months | Two months
  Moods and Feelings Questionnaire (Angold, 1995; Larson, Ingul, Jozefiak, Leikanger & Sund, 2016; Lundervold, Brevik, Possserud, Stormark & Hysing, 2013). Screen for Child Anxiety Related Disorders (Birmaher, Khetarpal, Cully, Brent &McKenzie, 1996)
Change from baseline internalized problems at one year | Two months
  Moods and Feelings Questionnaire (Angold, 1995; Larson, Ingul, Jozefiak, Leikanger & Sund, 2016; Lundervold, Brevik, Possserud, Stormark & Hysing, 2013). Screen for Child Anxiety Related Disorders (Birmaher, Khetarpal, Cully, Brent &McKenzie, 1996)
Baseline externalized problems | Two months
  Bullying (Olweus & Endresen, 1998) and The Bergen Questionnaire on Antisocial Behaviour (Bendixen & Olweus, 1999; Bendixen, Endresen & Olweus, 2003)
Change from externalized problems at eight months | Two months
  Bullying (Olweus & Endresen, 1998) and The Bergen Questionnaire on Antisocial Behaviour (Bendixen & Olweus, 1999; Bendixen, Endresen & Olweus, 2003)
Change from externalized problems at one year | Two months
  Bullying (Olweus & Endresen, 1998) and The Bergen Questionnaire on Antisocial Behaviour (Bendixen & Olweus, 1999; Bendixen, Endresen & Olweus, 2003)
Baseline teachers' reactions to sexual and gendered harassment (Teacher questionnaire) | Two months
  Modified versions of the primary outcome measures, including teachers' action, intentions to act and attitudes towards sexual and gendered harassment
Change from teachers' reactions to sexual and gendered harassment at eight months (Teacher questionnaire) | Two months
  Modified versions of the primary outcome measures, including teachers' action, intentions to act and attitudes towards sexual and gendered harassment
Change from teachers' reactions to sexual and gendered harassment at one year (Teacher questionnaire) | Two months
  Modified versions of the primary outcome measures, including teachers' action, intentions to act and attitudes towards sexual and gendered harassment

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Slaatten, Ph.D, Principal Investigator — NORCE Norwegian Research Centre AS
Locations (1):
- NORCE Norwegian Research Centre, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slaatten H, Haugland BSM, Bjorknes R, Fyhn T, Tveito TH, Poteat VP, Breivik K. Stop Sexual Harassment: A study protocol for a cluster randomised controlled trial in secondary schools in Norway. Front Public Health. 2023 Jan 9;10:1051983. doi: 10.3389/fpubh.2022.1051983. eCollection 2022. PMID 36699896